CLINICAL TRIAL: NCT01672957
Title: Non-interventional Clinical Study With Target of Kidney Function Follow-up in Routine Clinical Practice on De Novo Kidney Transplant Recipients Who Are on CellCept Immunosuppressive Combination Therapy in Routine Clinical Practice
Brief Title: An Observational Study on Renal Function in Kidney Transplant Participants on Immunosuppressive Therapy Containing Mycophenolate Mofetil
Acronym: ORANGE
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML27844
Record Dates: First submitted 2012-08-22; First posted 2012-08-27 (Estimated); Results first posted 2016-10-11 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-08

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — Mycophenolic Acid; Immunosuppression Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Renal Transplant Participants: Renal transplant participants who will be subjected to a combined immunosuppressive treatment containing mycophenolate mofetil, will be followed-up until the end of the study (after 12 months), or until the participant's death, withdrawal, or lost contact with the participant, whichever occurs first. The choice of treatment will be made prior to enrolment by the treating physician. The treatment will be administered according to applicable therapeutic protocol and Summary of Product Characteristics (SmPC).
  Interventions: Drug: Mycophenolate Mofetil; Drug: Immunosuppressive Therapy

INTERVENTIONS:
Drug: Mycophenolate Mofetil — Protocol does not specify any regimen for treatment. The choice of treatment will be made prior to enrollment by the treating physician.
  Other Names: CellCept
Drug: Immunosuppressive Therapy — Protocol does not specify any particular immunosuppressive drug and regimen for treatment. The choice of immunosuppressive therapy will be made prior to enrollment by the treating physician.

SUMMARY:
This observational study will evaluate renal function in participants who underwent renal allograft transplantation and are started on combined immunosuppressive treatment containing mycophenolate mofetil (CellCept). Eligible participants will be followed for 12 months following transplantation.

DETAILED DESCRIPTION:
The participant sampling method used in the Orange study was consecutive sampling, a non-probability sampling method where each participant meeting the study's inclusion and exclusion criteria is selected and enrolled in the study until the pre-set sample size is achieved.

Thus, in the Orange study de novo kidney transplanted participants, who were on mycophenolate mofetil immunosuppressive combination therapy in routine clinical practice, were selected in a consecutive manner (a non-probability sampling method) if they met the inclusion/exclusion criteria until 128 participants were recruited to the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants who underwent renal allograft transplantation and are started on combined immunosuppressive treatment containing mycophenolate mofetil in accordance with the indication provided by the SmPC of mycophenolate mofetil
* Date of study enrollment is the date of kidney transplantation

Exclusion Criteria:

* Contraindication included in the SmPC for capecitabine (Xeloda) prevailed, like: Hypersensitivity to active ingredient or any of the excipients of the product; Pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Renal allograft transplant participants initiated on combined immunosuppressive treatment containing mycophenolate mofetil
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2011-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- Hungary (2):
  - Budapest
  - Pécs

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: If Informed Consent Form (ICF) was signed after the transplantation, it was considered as a major protocol violation and reported separately from protocol violation in Participant Flow.
Groups:
- Renal Transplant Participants: Renal transplant participants who were subjected to a combined immunosuppressive treatment containing mycophenolate mofetil (CellCept), were followed-up until the end of the study (after 12 months), or until the participant's death, withdrawal, or lost contact with the participant, whichever occurred first. The choice of treatment was made prior to enrollment by the treating physician. The treatment was administered according to applicable therapeutic protocol and Summary of Product Characteristics (SmPC). The study protocol did not specify any treatment regimen.
Period: Overall Study
Arm/Group | Renal Transplant Participants
Started | 128
Intent-to-treat (ITT) Population | 123 (All enrolled participants who had no major protocol violation.)
Completed | 73
Not Completed | 55
Not completed — Protocol Violation | 48
Not completed — Death | 2
Not completed — ICF Signed After Transplantation | 5

BASELINE CHARACTERISTICS:
Population: ITT population included all enrolled renal transplant participants who received mycophenolate mofetil containing immunosuppressive combination therapy and had no major protocol violation.
Groups:
- Renal Transplant Participants: Renal transplant participants who were subjected to a combined immunosuppressive treatment containing mycophenolate mofetil, were followed-up until the end of the study (after 12 months), or until the participant's death, withdrawal, or lost contact with the participant, whichever occurred first. The choice of treatment was made prior to enrollment by the treating physician. The treatment was administered according to applicable therapeutic protocol and SmPC. The study protocol did not specify any treatment regimen.
Arm/Group | Renal Transplant Participants
Number analyzed (Participants) | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.60 (13.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 79

OUTCOME MEASURES:

1. Primary Outcome: Creatinine Clearance at 1 Month After Transplantation
Description: Creatinine clearance is an indicator of renal function. Creatinine clearance is the volume of blood plasma that is cleared of creatinine by the kidneys per unit time. Normal values for healthy, young males are in the range of 100-135 milliliters per minute (mL/min) and for females, 90-125 mL/min. Creatinine clearance decreases with age. A low creatinine clearance rate indicates poor kidney function.
Time Frame: Month 1
Population: ITT population. Number of participants analyzed = participants evaluable for creatinine clearance at specified time-point.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Renal Transplant Participants
Number analyzed (Participants) | 107
mL/min | 65.82 (18.32)

2. Primary Outcome: Creatinine Clearance at Month 6 After Transplantation
Description: Creatinine clearance is an indicator of renal function. Creatinine clearance is the volume of blood plasma that is cleared of creatinine by the kidneys per unit time. Normal values for healthy, young males are in the range of 100-135 mL/min and for females, 90-125 mL/min. Creatinine clearance decreases with age. A low creatinine clearance rate indicates poor kidney function.
Time Frame: Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Renal Transplant Participants
Number analyzed (Participants) | 76
mL/min | 73.38 (19.43)

3. Primary Outcome: Creatinine Clearance at Month 12 After Transplantation
Description: as for outcome 2
Time Frame: Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Renal Transplant Participants
Number analyzed (Participants) | 70
mL/min | 69.69 (21.05)

4. Primary Outcome: Glomerular Filtration Rate (GFR) at Month 1 After Transplantation
Description: GFR is an index of kidney function. GFR describes the flow rate of filtered fluid through the kidney. A normal GFR is greater than (>) 90 mL/min, although children and older people usually have a lower GFR. Lower values indicates poor kidney function. A GFR less than (<) 15 mL/min indicates kidney failure.
Time Frame: Month 1
Population: ITT population. Number of participants analyzed = participants evaluable for GFR at specified time-point.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Renal Transplant Participants
Number analyzed (Participants) | 118
mL/min | 53.54 (33.43)

5. Primary Outcome: GFR at Month 6 After Transplantation
Description: GFR is an index of kidney function. GFR describes the flow rate of filtered fluid through the kidney. A normal GFR is > 90 mL/min, although children and older people usually have a lower GFR. Lower values indicates poor kidney function. A GFR < 15 mL/min indicates kidney failure.
Time Frame: Month 6
Population: ITT population. Number of participants analyzed = participants evaluable for GFR at specified time-point.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Renal Transplant Participants
Number analyzed (Participants) | 83
mL/min | 56.78 (15.36)

6. Primary Outcome: GFR at Month 12 After Transplantation
Description: as for outcome 5
Time Frame: Month 12
Population: ITT population. Number of participants analyzed = participants evaluable for GFR at specified time-point.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Renal Transplant Participants
Number analyzed (Participants) | 65
mL/min | 58.03 (16.29)

7. Secondary Outcome: Mean Dose of Mycophenolate Mofetil
Time Frame: Baseline, Months 1, 6, and 12
Population: ITT population. Number of participants analyzed = participants evaluable for this outcome measure. Here 'n' signifies number of participants evaluable at specified time-points.
Measure: Mean (Standard Deviation); unit: milligrams (mg)
Arm/Group | Renal Transplant Participants
Number analyzed (Participants) | 121
milligrams (mg)
  Baseline (n=121) | 2033.06 (357.86)
  Month 1 (n=119) | 1718.49 (543.21)
  Month 6 (n=88) | 1457.39 (754.51)
  Month 12 (n=69) | 1539.86 (669.21)

8. Secondary Outcome: Percentage of Participants Who Received Other Immunosuppressive Agents in Combination With Mycophenolate Mofetil
Description: Participants could have received more than one other immunosuppressive agents, at the discretion of treating physician. Percentage of participants who received 1 other immunosuppressive agent, 2 other immunosuppressive agents, and 3 other immunosuppressive agents are reported.
Time Frame: Baseline, Months 1, 6, and 12
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Renal Transplant Participants
Number analyzed (Participants) | 121
percentage of participants
  1 Other agent: at baseline (n=121) | 0.8
  1 Other agent: at Month 1 (n=119) | 0.8
  1 Other agent: at Month 6 (n=86) | 2.3
  1 Other agent: at Month 12 (n=69) | 7.2
  2 Other agents: at baseline (n=121) | 90.9
  2 Other agents: at Month 1 (n=119) | 99.2
  2 Other agents: at Month 6 (n=86) | 97.7
  2 Other agents: at Month 12 (n=69) | 92.8
  3 Other agents: at baseline (n=121) | 8.3
  3 Other agents: at Month 1 (n=119) | 0
  3 Other agents: at Month 6 (n=86) | 0
  3 Other agents: at Month 12 (n=69) | 0

9. Secondary Outcome: Percentage of Participants With Acute Rejection
Description: Percentage of participants who experienced acute rejection within 1 month of transplantation, Month 2 to Month 6 after transplantation, Month 7 to Month 12 after transplantation are reported.
Time Frame: Baseline to Month 1, Months 2 to 6, Months 7 to 12
Population: Safety population included all enrolled renal transplant participants who received mycophenolate mofetil containing immunosuppressive combination therapy (safety population=128). Number of participants analyzed = participants evaluable for this outcome measure. Here 'n' signifies number of participants evaluable at specified time-points.
Measure: Number; unit: percentage of participants
Arm/Group | Renal Transplant Participants
Number analyzed (Participants) | 127
percentage of participants
  Baseline to Month 1 (n=127) | 16.5
  Months 2 to 6 (n=124) | 0.8
  Months 7 to 12 (n=111) | 0.9

10. Secondary Outcome: Percentage of Participants With Graft Survival
Description: Graft survival was defined as those participants who did not experience graft loss. Graft loss defined as physical loss (nephrectomy), functional loss (necessitating maintenance dialysis for >8 weeks), re-transplant or death during the first 12 months after transplantation.
Time Frame: Months 1, 6, and 12
Population: Safety population. Number of participants analyzed = participants evaluable for this outcome measure. Here 'n' signifies number of participants evaluable at specified time-points.
Measure: Number; unit: percentage of participants
Arm/Group | Renal Transplant Participants
Number analyzed (Participants) | 127
percentage of participants
  Month 1 (n=127) | 100
  Month 6 (n=123) | 99.2
  Month 12 (n=111) | 98.4

ADVERSE EVENTS:
Time Frame: From Baseline up to Month 12
Description: Safety population.
Arm/Group | Renal Transplant Participants
Serious Adverse Events (participants affected / at risk) | 33/128
Other Adverse Events (participants affected / at risk) | 51/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Renal Transplant Participants (N=128)
Acute myocardial infarction (Cardiac disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Sudden death (General disorders) | 1
Kidney transplant rejection (Immune system disorders) | 4
Transplant rejection (Immune system disorders) | 14
Cystitis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Postoperative abscess (Infections and infestations) | 1
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 1
Perirenal haematoma (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2
Ureteric anastomosis complication (Injury, poisoning and procedural complications) | 2
Blood creatinine increased (Investigations) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Pyelocaliectasis (Renal and urinary disorders) | 2
Tubulointerstitial nephritis (Renal and urinary disorders) | 1
Ureteral disorder (Renal and urinary disorders) | 1
Ureterolithiasis (Renal and urinary disorders) | 1
Varicocele (Reproductive system and breast disorders) | 1
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 1
Haematoma (Vascular disorders) | 2
Urinary tract infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Renal Transplant Participants (N=128)
Diarrhoea (Gastrointestinal disorders) | 19
Hyperuricaemia (Renal and urinary disorders) | 7
Urinary tract infection (Renal and urinary disorders) | 24
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 10
Anemia (Blood and lymphatic system disorders) | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.